CLINICAL TRIAL: NCT03503058
Title: Safety, Tolerability, Immunogenicity and Protective Efficacy Against Naturally-Transmitted Malaria in Eastern Indonesia of Two Plasmodium Falciparum Sporozoite Vaccines, Sanaria® PfSPZ Vaccine and Sanaria® PfSPZ-CVac: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Trial in Healthy Indonesian Adults
Brief Title: Safety, Tolerability, Immunogenicity and Protective Efficacy of PfSPZ Vaccine and PfSPZ-CVac in Indonesian Adults Against Naturally-Transmitted Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Oxford University Clinical Research Unit Indonesia (Other); Indonesia University (Other); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IDSPZV1
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; Sporozoites; PfSPZ
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Chemoprevention; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): N=124 will receive PfSPZ Vaccine; three doses of 9x10^5 PfSPZ of PfSPZ Vaccine administered by direct venous inoculation (DVI) given on day 1, 8 and 29.
  Interventions: Biological: PfSPZ Vaccine
- Group 2 (Placebo Comparator): N=62 will receive normal saline; three doses of NS administered by DVI given on day 1, 8 and 29.
  Interventions: Other: Normal Saline
- Group 3 (Experimental): N=124 will receive PfSPZ Challenge under chloroquine (CQ) chemoprophylaxis; three doses of 2x10^5 PfSPZ of PfSPZ Challenge administered by DVI on day 1, 29 and 57, with weekly CQ.
  Loading Dose: 10 mg/kg of CQ base (will be orally administered as a single loading dose to the participant by the study staff via directly observed therapy on PfSPZ-CVac Day -2.
  Weekly Dose: Subsequent doses of maintenance dose CQ (5 mg/kg CQ base) will be given weekly as a single dose, with the last dose 5 days after the last dose of PfSPZ Challenge.
  Interventions: Biological: PfSPZ Challenge under chloroquine (CQ) chemoprophylaxis
- Group 4 (Placebo Comparator): N=62 will receive normal; three doses of NS administered by DVI given on day 1, 29 and 57, with weekly CQ.
  Loading Dose: 10 mg/kg of CQ base (will be orally administered as a single loading dose to the participant by the study staff via directly observed therapy on PfSPZ-CVac Day -2.
  Weekly Dose: Subsequent doses of maintenance dose CQ (5 mg/kg CQ base) will be given weekly as a single dose, with the last dose 5 days after the last dose of PfSPZ Challenge.
  Interventions: Other: Normal Saline; Drug: Chloroquine chemoprophylaxis alone

INTERVENTIONS:
Biological: PfSPZ Vaccine — Radiation-attenuated, aseptic, purified, cryopreserved Plasmodium falciparum sporozoites (PfSPZ Vaccine)
  Arms: Group 1
Biological: PfSPZ Challenge under chloroquine (CQ) chemoprophylaxis — Infectious, aseptic, purified, cryopreserved Plasmodium falciparum sporozoites (PfSPZ Challenge) administered under CQ chemoprophylaxis
  Loading Dose: 10 mg/kg of CQ base (will be orally administered as a single loading dose to the participant by the study staff via directly observed therapy on PfSPZ-CVac Day -2.
  Weekly Dose: Subsequent doses of maintenance dose CQ (5 mg/kg CQ base) will be given weekly as a single dose, with the last dose 5 days after the last dose of PfSPZ Challenge.
  Other Names: PfSPZ-CVac
  Arms: Group 3
Other: Normal Saline — 0.9% Sodium chloride
  Other Names: NS
  Arms: Group 2; Group 4
Drug: Chloroquine chemoprophylaxis alone — Loading Dose: 10 mg/kg of CQ base (will be orally administered as a single loading dose to the participant by the study staff via directly observed therapy on NS Day -2.
  Weekly Dose: Subsequent doses of maintenance dose CQ (5 mg/kg CQ base) will be given weekly as a single dose, with the last dose 5 days after the last dose of NS.
  Other Names: CQ
  Arms: Group 4

SUMMARY:
The study is a double-blind, randomized, placebo-controlled, Phase 2 clinical trial that will assess the safety, tolerability, immunogenicity and protective efficacy of PfSPZ Vaccine and PfSPZ-CVac against naturally occurring malaria in healthy Indonesian soldiers deployed to eastern Indonesia.

DETAILED DESCRIPTION:
The study is a double-blind, randomized, placebo-controlled, Phase 2 clinical trial that will assess the safety, tolerability, immunogenicity and protective efficacy of PfSPZ Vaccine and PfSPZ-CVac against naturally occurring malaria in 372 healthy Indonesian soldiers aged 18-55 years who will be deployed in malarious eastern Indonesia.

PfSPZ Vaccine and PfSPZ-CVac:

Participants will be randomized to immunization with three doses of PfSPZ Vaccine (Group 1), normal saline (NS) placebo (Group 2) and PfSPZ-CVac (PfSPZ Challenge + CQ) (Group 3) or NS placebo + CQ (Group 4); randomization to four groups will be 1 : 0.5 : 1 : 0.5.

The study has three phases: immunization and follow-up at the home base; deployment to eastern Indonesia for 6 to 9 months (surveillance period #1); redeployment to the home base for 6 months (surveillance period #2); study participation will be up to 20 months per participant, and the entire clinical trial will last approximately 28 months if deployment lasts 9 months. A research monitor (RM) (= medical monitor = safety monitor) and a safety monitoring committee (SMC) will provide safety oversight. External study monitoring will be the responsibility of Sanaria or Sanaria's designated and authorized representative in Indonesia. Screening will be done within 56 days of enrollment and immunizations will be completed prior to deployment. Screening evaluation includes an electrocardiogram (ECG) performed at screening. Subjects with clinically significant abnormal cardiovascular symptoms or findings will be excluded and referred to a cardiologist for further evaluation; individuals with a history of non-febrile seizures will also be excluded. Solicited adverse events will be monitored for 7 days after each PfSPZ Vaccine/placebo administration and for 14 days after each PfSPZ-CVac/placebo administration; unsolicited adverse events will be followed during the immunization period and up to 2 weeks after the last immunization if the deployment schedule allows; serious adverse events (SAEs) will be monitored throughout the study. Follow-up of AEs occurs until resolution or stability. Case report forms (CRFs) will serve as the repository of source documents and other relevant data for each study subject. Only information that cannot be collected initially into the CRF (namely, laboratory test results, ECGs and adverse event (AE) medical records, etc.) will first be collected onto separate source documents before transcription into the CRF. The information in the CRF will then be manually entered directly into the internet data system by independent data entry technicians.

Study Arms:

Group 1 (n=124): Three doses of 9x10^5 PfSPZ of PfSPZ Vaccine. Group 2 (n=62): Three doses of NS. Group 3 (n=124): Three doses of 2x10^5 PfSPZ of PfSPZ Challenge and weekly CQ. Group 4 (n=62): Three doses of NS and weekly CQ.

ELIGIBILITY:
Inclusion Criteria:

* A male aged 18-55 years at the time of screening.
* Assigned to the battalion of study and programmed to accompany it to eastern Indonesia for the duration of the deployment.
* Freely provides written informed consent to participate in the study.
* Agrees to adhere to Indonesian military medical guidance regarding screening and treatment of malaria.
* Physical examination and laboratory results without clinically significant findings that would jeopardize the safety of the participant or the integrity of the study, and a body mass index (BMI) ≤35 kg/m^2.

Exclusion Criteria:

* Previous vaccination with an investigational malaria vaccine.
* Use of an investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days before the first study vaccination, or planned use up to 30 days after last vaccination.
* Chronic administration (defined as more than 14 days) of immunosuppressant or other immune-modifying drugs within six months before the first vaccination. This includes any dose level of oral steroids, but not inhaled steroids or topical steroids.
* Administration or planned administration of 1 live or 3 or more other type vaccines in the period beginning 28 days before the first study vaccination and ending 28 days after the last vaccination.
* Confirmed or suspected immunosuppressive or immunodeficient condition.
* Confirmed or suspected autoimmune disease.
* History of allergic reactions or anaphylaxis to CQ or other 4-aminoquinolone derivatives.
* History of serious allergic reactions to a drug (anaphylaxis, or requiring hospitalization).
* History of allergy to phosphate buffered saline or human serum albumin.
* Use or planned use of any drug with anti-malarial activity during the course of the study except for antimalarial medication administered by study clinicians.
* History of splenectomy.
* Laboratory evidence of liver disease (the final decision will be made by the PI and clinical officers, but in general a volunteer will be excluded if any of the screening liver function tests (ALT, bilirubin, gamma GTP) are > double the upper limit of normal measured twice without an explanation for the abnormal values).
* Laboratory evidence of renal disease (serum creatinine > 1.5 mg/dL. measured twice).
* Laboratory evidence of hematologic disease (platelet count or hemoglobin <80% of the lower limit of normal for Indonesia measured twice).
* Abnormal screening ECG showing prolonged QTc interval (>450 msec) or any signs of arrythmia/irregularity, ischemia, cardiac enlargement considered considered indicative of acute or chronic cardiovascular disease.
* Acute or chronic pulmonary, cardiovascular, hepatic, renal or neurological condition, severe malnutrition, or any other clinical findings that may increase the risk of participating in the study as determined by the principal investigator or her designee.
* Administration of immunoglobulin and/or any blood products within the three months preceding the first study vaccination or planned administration during the study period.
* Simultaneous participation in any other interventional clinical trial.
* Other conditions that in the opinion of the principal investigator or her designee would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol or might compromise the integrity of the data.
* Any evidence of active malaria, whether symptomatic or asymptomatic, confirmed by RDT, microscopy or PCR before first injection of PfSPZ Vaccine or PfSPZ-CVac, unless treated by the clinical team.
* History of non-febrile seizures or atypical febrile seizures.
* Under treatment for tuberculosis.
* Laboratory evidence of active infection with hepatitis B, or hepatitis C.
* Subjects with > 10% 5-year cardiovascular risk (fatal and non-fatal) based on the Gaziano scoring system; subjects in the 18-34 year old age group will be assessed as though they are in the 35-44 age group.
* History of psychiatric disorders (such as personality disorders, anxiety disorders, or schizophrenia) or behavioral tendencies (including active alcohol or drug abuse) discovered during the screening process that in the opinion of the investigator would make compliance with the protocol difficult.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 345 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
The number of adverse events occurring after investigational product (IP) administration | a. 7 days (PfSPZ Vaccine) or 12 (first two doses) or 14 (third dose) days (PfSPZ-CVac) of each administration. b. From day of immunization until end of study (24 months). c. 14 days of each administration
  a. The proportion of participants experiencing of solicited AEs occurring within 7 days (PfSPZ Vaccine) or 14 days (PfSPZ-CVac) of each administration of investigational product (IP).
  b) The proportion of participants experiencing serious adverse events (SAEs) deemed related to IP during active participation in the trial.
  c) The proportion of participants experiencing unsolicited AEs occurring within 14 days of each administration of IP deemed related to vaccination or placebo administration.
The number of confirmed first infections with Pf | 10 days after arriving in eastern Indonesia through 10 days after leaving eastern Indonesia.
  The number of confirmed first clinical malaria cases caused by Pf among subjects receiving vaccine vs. placebo during the period from 10 days after arriving in eastern Indonesia through 10 days after leaving eastern Indonesia.

SECONDARY OUTCOMES:
The number of confirmed first infections* caused by Pf | 10 days after arriving in eastern Indonesia through 10 days after leaving eastern Indonesia
  The number of confirmed first infections* caused by Pf among subjects receiving vaccine vs. placebo during the period from 10 days after arriving in eastern Indonesia through 10 days after leaving eastern Indonesia.
  * thick blood smears from asymptomatic individuals will be read retrospectively, so there is no interference in ascertaining the number of clinical cases, which is the primary VE endpoint.
The number of confirmed first clinical malaria cases caused by Pv | 10 days after arriving in eastern Indonesia through 10 days after leaving eastern Indonesia.
  The number of confirmed first clinical malaria cases caused by Pv among subjects receiving vaccine vs. placebo during the period from 10 days after arriving in eastern Indonesia through 10 days after leaving eastern Indonesia.
The number of confirmed first infections with Pv in eastern Indonesia | 10 days after arriving in eastern Indonesia through 10 days after leaving eastern Indonesia.
  The number of confirmed first infections* caused by Pv among subjects receiving vaccine vs. placebo during the period from 10 days after arriving in eastern Indonesia through 10 days after leaving eastern Indonesia.
  * thick blood smears from asymptomatic individuals will be read retrospectively, so there is no interference in ascertaining the number of clinical cases, which is the primary VE endpoint.
The number of confirmed relapsing infections from Pv | 10 days after arriving in eastern Indonesia through 10 days after leaving eastern Indonesia.
  The number of confirmed relapsing infections from latent liver stages of Pv identified post-exposure in a malaria-free area.
Humoral immune responses | 14 days after the third dose of vaccine
  The humoral immune responses* induced by vaccination compared to those induced by placebo administration comparing vaccinees to controls; (b) the association between the immune responses and protection (no parasitemia or clinical malaria occurring during surveillance).
  *(i) Levels of antibodies against Pf circumsporozoite protein (CSP) by ELISA 2 weeks after the third dose of vaccine; (ii) Optional: Levels of antibodies against PvCSP by ELISA 2 weeks after the third dose of vaccine; (iii) Optional: Levels of antibodies against other Pf and Pv proteins, PfSPZ, PvSPZ and Pf and Pv asexual erythrocytic stages (AES) 2 weeks after the third dose; (iv) Optional: inhibition of sporozoite invasion assay,

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Baird, Ph.D., Study Director — Eijkman-Oxford Clinical Research Unit, Eijkman Institute of Molecular Biology, Indonesia; Erni J Nelwan, MD, Ph.D., Principal Investigator — Department of Internal Medicine, Universitas Indonesia
Locations (2):
- Indonesia (2):
  - Department of Internal Medicine, Universitas Indonesia, Jakarta
  - Eijkman-Oxford Clinical Research Unit, Eijkman Institute of Molecular Biology, Jakarta